CLINICAL TRIAL: NCT04157816
Title: Digital Compared to Conventional Training for Non-Specialist Health Workers to Deliver a Brief Psychological Treatment for Depression in Primary Care in India: A Three-Arm Randomized Controlled Trial
Brief Title: Digital Training for Non-Specialist Health Workers to Deliver a Brief Psychological Treatment for Depression
Acronym: ESSENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Sangath (Other)
Responsible Party: Principal Investigator, Vikram Patel, Professor of Global Health and Social Medicine, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: U19MH113211-03 (NIH)
Record Dates: First submitted 2019-11-03; First posted 2019-11-08 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Depression; Mental Disorder; Psychological
Keywords: health worker training; non-specialist health worker; community health worker; task sharing; common mental disorders; low-resource setting; primary care; global mental health; digital technology; mobile health
MeSH Terms: conditions — Depression; Mental Disorders

STUDY DESIGN:
Intervention Model Description: This study employs a 3-arm parallel randomized controlled trial design. Participants are randomly allocated to one of three training interventions: 1) low-intensity digital training (DGT); 2) high-intensity digital training with additional coaching support (DGT+); and 3) traditional face-to-face training (F2F).
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this trial, the Outcome Assessors administering study assessments at baseline and at endpoint will be masked to the intervention arm that participants are allocated to receive. The Study Investigators will also be masked to the intervention arm that participants are allocated to receive. Masking Outcome Assessors and Study Investigators will minimize potential bias due to knowledge of which arm the participant is allocated to, and can ensure unbiased ascertainment of study outcomes is possible. For allocation concealment, the intervention allocation for each participant will not be revealed to the participant until they have been enrolled into the trial, to avoid selection bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital Training (DGT) (Experimental): Participants allocated to this arm receive a low-intensity digital program accessible by smart phone app for training non-specialist health workers to deliver an evidence-based brief psychological treatment for depression, called the Healthy Activity Program (HAP), in primary care settings in India.
  Interventions: Other: Digital Training
- Digital Training with Coaching Support (DGT+) (Experimental): Participants allocated to this arm receive a high-intensity digital program accessible by smart phone app augmented with weekly telephone coaching support for training non-specialist health workers to deliver an evidence-based brief psychological treatment for depression, called the Healthy Activity Program (HAP), in primary care settings in India.
  Interventions: Other: Digital Training; Other: Coaching Support
- Face-to-Face Training (Active Comparator): Participants allocated to this arm receive a traditional classroom-based (face-to-face) program hosted in community settings for training non-specialist health workers to deliver an evidence-based brief psychological treatment for depression, called the Healthy Activity Program (HAP), in primary care settings in India.
  Interventions: Other: Face-to-Face Training

INTERVENTIONS:
Other: Face-to-Face Training — This intervention is a traditional classroom-based (face-to-face) training program for non-specialist health workers offering instruction for the delivery of the Healthy Activity Program (HAP) in primary care settings. HAP is an evidence-based brief psychological treatment for depression. The classroom instruction follows the HAP manuals and is facilitated by an experienced counselor with certification as a Master Trainer, meaning that they have significant experience delivering HAP to patients with depression in clinical settings and also training other health workers in the delivery HAP. The total duration of classroom instruction is 6 days.
  Arms: Face-to-Face Training
Other: Digital Training — This 4-week digital training program for non-specialist health workers is accessed through a smart phone app and offers instruction in the delivery of the Healthy Activity Program (HAP) in primary care settings. HAP is an evidence-based brief psychological treatment for depression. The digital training covers the same content as the Face-to-Face training. The course includes 16 modules with video lectures, role-play videos, graphics, slide presentations, quizzes, and assessment questions. Participants also receive low-intensity support to enhance their learning experience and sustain engagement, including: 1) access to an automated 'Help Line' that participants can call any time with questions about the program; 2) weekly automated messages sent through the mobile app to encourage participants; and 3) automated messages and phone calls to participants who show prolonged periods of inactivity in the mobile app to offer technical support and help them complete the training program.
  Arms: Digital Training (DGT); Digital Training with Coaching Support (DGT+)
Other: Coaching Support — Individualized remote coaching is a form of high-intensity support that will be used to help sustain participant engagement in the digital training program and promote success in progressing through the course. Each week, a Coach will phone participants and offer encouragement and support related to the course. The phone call will last no more than 60 minutes. The Coach will be someone who has successfully completed the course, and therefore can offer first hand knowledge of the content. During the coaching session, the coach will review the participants' progress through the course, offer praise and encouragement, discuss any challenges or questions related to the course content, and review the participants' goals and plans for the upcoming week. Each participant will receive a maximum of 4 remote coaching sessions (1 per week over the 4-week training program).
  Arms: Digital Training with Coaching Support (DGT+)

SUMMARY:
The purpose of this 3-arm randomized controlled trial is to compare two forms of digital training (i.e., low-intensity and high-intensity) with traditional face-to-face training of non-specialist health workers to deliver an evidence-based brief psychological treatment for depression called the Healthy Activity Program (HAP) in primary care settings in India. This study will evaluate a low-intensity digital training program (DGT) compared with traditional face-to-face training (F2F) on change in competence outcomes and cost-effectiveness. This study will also evaluate a high-intensity digital training program with the addition of individualized coaching support (DGT+) compared with traditional F2F on change in competence outcomes and cost-effectiveness.

DETAILED DESCRIPTION:
Few individuals living with depression in India have access to adequate treatment in primary care settings. Task-sharing, which involves building capacity of frontline non-specialist health workers to deliver evidence-based treatment for common mental disorders such as depression, is an effective approach for bridging these gaps in available care. This emphasizes the need for novel approaches to scale up training efforts and to support the development of a skilled and competent workforce capable of delivering high quality treatment for depression in primary care settings. Therefore, the purpose of this study is to compare two forms of digital training (i.e., low-intensity and high-intensity) with traditional face-to-face training of non-specialist health workers to deliver an evidence-based brief psychological treatment for depression called the Healthy Activity Program (HAP) in primary care settings in India. This trial uses a 3-arm randomized controlled design. This study will evaluate a low-intensity digital training (DGT) compared with traditional face-to-face training (F2F) on change in competence outcomes and cost-effectiveness; and evaluate a high-intensity digital training with the addition of individualized coaching support (DGT+) compared with traditional F2F on change in competence outcomes and cost-effectiveness. In this trial, a total of 336 non-specialist health workers will be recruited from community health centers in Sehore District of Madhya Pradesh, a large and predominantly rural state situated in central India. This trial will generate knowledge on the most effective and cost-effective approaches to address the critical knowledge gap regarding the training of non-specialist health workers to deliver an evidence-based brief psychological treatment for depression in a low-resource setting. The findings from this trial will inform broader efforts to develop a mental health workforce necessary for scaling up brief psychological therapies for common mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years)
* Non-specialist health worker
* Minimum education level 8th Standard
* Willingness to complete training to deliver HAP
* Willingness to stay in the study area during the trial period

Exclusion Criteria:

* Significant speech, sight, or hearing impairment
* Illiterate/ who cannot read and write
* Prior participation in the formative research and pilot testing (during the development of the training programs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Competency | Change from Baseline to up to 8 weeks.
  26-item multiple choice exam to assess the competency of the non-specialist health workers in delivering the Healthy Activity Program (HAP) after training. The measure consists of clinical vignettes followed by multiple-choice questions focused predominantly on assessing applied knowledge. Scores on the measure range from 0 to 26, with higher scores indicating higher levels of competency for delivering HAP. There are three different equivalent versions of this 26-item measure, and each participant will be assessed randomly with one of these at each of the two time points, ensuring that the same test is not used twice.To assess change in competency between two time points, this measure will be collected at baseline and at up to 8 weeks.

SECONDARY OUTCOMES:
Change in Mental Health Knowledge, Attitude, and Behavior | Change from Baseline to up to 8 weeks.
  13-item self-report questionnaire uses a 5-point Likert scale to ascertain non-specialist health workers' knowledge, attitudes, and behavior about different aspects of mental health. Scores range from 13 to 65, with higher scores indicating greater knowledge and better attitudes and behaviors towards persons living with a mental illness. Lower scores on this measure suggest lower levels of knowledge and greater stigma towards mental illness. This is important to measure because completion of the training program may contribute to improvements in knowledge, attitudes and behaviors about mental health. To assess change in mental health knowledge, attitudes, and behavior between two time points, this measure will be collected at baseline and at up to 8 weeks.

OTHER OUTCOMES:
Costs Incurred During Participation in the Training Program | Up to 8 weeks.
  The direct and indirect costs incurred by participants while completing each of the training programs will be collected after completion of the training program at up to 8 weeks. Participants will complete an 8-item questionnaire about the time, travel, and any monetary costs incurred during their completion of the training program. This questionnaire is not scored on a scale; each item will be examined as it relates to specific details about costs related to participation in the training program.
Satisfaction with the Training Program | Up to 8 weeks.
  This 26-item questionnaire assesses participants' satisfaction with the training programs (either of the two forms of digital training or the traditional Face-to-Face training). This satisfaction questionnaire will be collected after completion of the training program at up to 8 weeks. Each of the 26-items on the questionnaire is rated on a 6-point Likert scale. The items cover feasibility, acceptability, adoption, and appropriateness of the training program. Scores on this questionnaire range from 26 to 156, with higher scores indicating greater satisfaction with the training program. The purpose of the questionnaire is to identify strengths and weaknesses related to factors and program content that affect participants' motivation and engagement in the training program.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Patel, MD, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Sangath, Bhopal, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) from this trial will be shared with the scientific community according to the National Institute of Mental Health (NIMH) Data Archive Data Sharing terms and conditions. Data will have all direct or indirect identifiable information removed before being submitted to the NIMH Data Archive (NDA). After the trial, the investigators will send de-identified information from participants to NDA. Researchers can access this de-identified data by submitting a request to NIMH. Data sharing with NDA offers no direct benefit to participants, though the information provided to NDA may help researchers around the world treat future mental health challenges so that they have better outcomes. Study participants can choose not to have their de-identified data shared with NDA. These details about data sharing with NDA are described in the participant consent form, and additional information is available at the NDA website.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) will be submitted to the NIMH Data Archive within 12 months after completion of the trial according to the NDA submission schedule and policies.
Access Criteria: There is no plan to restrict access to anonymized data for research purposes. However, access will be provided through the NDA Data Access Committee (DAC). Investigators and institutions seeking data from NDA will be expected to meet data security measures and will be asked to submit a Data Use Certification.
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Patel V, Weobong B, Weiss HA, Anand A, Bhat B, Katti B, Dimidjian S, Araya R, Hollon SD, King M, Vijayakumar L, Park AL, McDaid D, Wilson T, Velleman R, Kirkwood BR, Fairburn CG. The Healthy Activity Program (HAP), a lay counsellor-delivered brief psychological treatment for severe depression, in primary care in India: a randomised controlled trial. Lancet. 2017 Jan 14;389(10065):176-185. doi: 10.1016/S0140-6736(16)31589-6. Epub 2016 Dec 15. PMID 27988143
- [Background] Muke SS, Shrivastava RD, Mitchell L, Khan A, Murhar V, Tugnawat D, Shidhaye R, Patel V, Naslund JA. Acceptability and feasibility of digital technology for training community health workers to deliver brief psychological treatment for depression in rural India. Asian J Psychiatr. 2019 Oct;45:99-106. doi: 10.1016/j.ajp.2019.09.006. Epub 2019 Sep 7. PMID 31557716
- [Background] Muke SS, Tugnawat D, Joshi U, Anand A, Khan A, Shrivastava R, Singh A, Restivo JL, Bhan A, Patel V, Naslund JA. Digital Training for Non-Specialist Health Workers to Deliver a Brief Psychological Treatment for Depression in Primary Care in India: Findings from a Randomized Pilot Study. Int J Environ Res Public Health. 2020 Sep 1;17(17):6368. doi: 10.3390/ijerph17176368. PMID 32883018
- [Background] Naslund JA, Tugnawat D, Anand A, Cooper Z, Dimidjian S, Fairburn CG, Hollon SD, Joshi U, Khan A, Lu C, Mitchell LM, Muke S, Nadkarni A, Ramaswamy R, Restivo JL, Shrivastava R, Singh A, Singla DR, Spiegelman D, Bhan A, Patel V. Digital training for non-specialist health workers to deliver a brief psychological treatment for depression in India: Protocol for a three-arm randomized controlled trial. Contemp Clin Trials. 2021 Mar;102:106267. doi: 10.1016/j.cct.2021.106267. Epub 2021 Jan 6. PMID 33421650
- [Derived] Joshi U, Haney JR, Sequeira M, Singla DR, Patel V, Bhan A, Cooper Z, Naslund JA. Adaptation and translation of a scalable measure for assessing health worker competence to deliver a brief psychological intervention: A case study from central India of its comparison to a performance-based measure. Psychiatr Q. 2023 Mar;94(1):33-47. doi: 10.1007/s11126-022-10007-6. Epub 2022 Dec 20. PMID 36536268